CLINICAL TRIAL: NCT03870932
Title: Effects of a Motor Imagery Exercise Protocol on Chronic Pain and Emotional Distress in Patients With Fibromyalgia: a Pilot Study
Brief Title: Effects of a Motor Imagery Exercise Protocol in Patients With Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Teresa Paolucci, Assistant Medical Director (Physiatrist), University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: URomLS-2018
Record Dates: First submitted 2019-03-10; First posted 2019-03-12 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Fibromyalgia; Pain, Chronic; Image, Body; Psychological Distress
Keywords: Fibromyalgia; Pain; Imagery
MeSH Terms: conditions — Fibromyalgia; Chronic Pain; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motor imagery rehabilitative group (MIG) (Experimental): All patients performed 10 treatment sessions, lasting 60 to 90 minutes, twice a week, in groups of three to four patients. The gold standard was to choose simple and safe exercises in order to encourage the patient to repeat the schedule at home. The exercises proposed in the MIG have been chosen respecting the following principles: slowness, painlessness, promoting attention, easy to imagine. The main purpose of motor imagery-based exercises was to bring the patient back to "feeling and self-perceiving" the execution of the movement. More than the "quantity" of repetition, the "quality" of the movement, free from pain, was important.
  Interventions: Other: Motor Imagery physical therapy
- Control rehabilitative Group (CG) (Active Comparator): The CG received a conventional rehabilitation protocol, based on ten 1-hour sessions, held twice a week (over a 5-week period), previously investigated as efficient in FM by the authors and published. The exercises included low-to-moderate impact aerobic training, walking in a circle, alternating with periods of going up and down the stairs (3 steps for 10 minutes), for a total of 20 consecutive minutes, posture exercises for the back and proprioceptive exercises for the trunk, to improve axial stability. Each exercise was repeated 10 times (3 sets of 10), with a resting period of at least 3 minutes between sets. All sessions ended with stretching and diaphragmatic breathing exercises.
  Interventions: Other: Conventional physical therapy

INTERVENTIONS:
Other: Motor Imagery physical therapy
  Arms: Motor imagery rehabilitative group (MIG)
Other: Conventional physical therapy
  Arms: Control rehabilitative Group (CG)

SUMMARY:
The aim of this study was to evaluate the efficacy of a novel approach with a motor imagery-based exercise program versus conventional rehabilitative approach in fibromyalgia syndrome (FM): reduction of pain was set as the primary outcome.

DETAILED DESCRIPTION:
Evidence about the therapeutic efficacy of exercise intervention programs in FM is still low and many authors suggested improving standardized exercise prescription for FM to achieve optimal results. In the literature, as an alternative approach, rehabilitative protocols in Group Music and Imagery seem to improve well-being and reduce anxiety in women with FM and suggest that Music and Imagery may help diminish pain intensity and depression. A rehabilitative approach should also consider the psychological and emotional aspects and, when possible, be accompanied by cognitive-behavioral therapy. The purpose of this research is to evaluate the possible efficacy of a novel approach with a motor imagery-based exercise program versus conventional rehabilitative approach in FM syndrome: the reduction of pain was set as the primary outcome as well as taking into account the patient's psychological and emotional condition. This study was designed as a double-blind, randomized, controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* experienced widespread pain for more than 3 months
* pain with 4 kg/cm2 pressure at 11 or more of the 18 tender points
* aged 18 to 60 years
* pharmacological therapeutic regimen must have been stable for at least three months before

Exclusion Criteria:

* pregnant women
* pacemaker wearers
* overlapping painful conditions
* presence of autoimmune or hematologic diseases
* psychiatric disorders in pharmacological and psychological treatment
* other causes of chronic pain
* other diseases such as epilepsy, tumors, major neurological problems and diabetes

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
Fibromyalgia Impact Questionnaire (FIQ) | 0-4-12 weeks
  self-administered instrument to assess the current health status of patients with fibromyalgia
Health Assessment Questionnaire (HAQ) | 0-4-12 weeks
  comprehensive measure of outcome in patients with a wide variety of chronic diseases
Fibromyalgia Assessment Status (FAS) | 0-4-12 weeks
  self-administered index that combines fatigue, sleep disturbances and pain in 16 non-articular sites
Visual Analogue Scale (VAS) | 0-4-12 weeks
  Instrument to assess unidimensional measure of pain intensity. VAS was presented in a coloured scale with a middle point, graduations and numbers. Under the scale there was a straight horizontal line of fixed length, 100 mm. The ends were defined as the limits of the parameter to be measured (pain in the last 24 hours), orientated from the left (worst, no pain) to the right (best, worst pain to be imagined). The score is determined by measuring the distance (cm) on the 10 cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-10.
Hamilton Anxiety Rating Scale (HAM-A) | 0-4-12 weeks
  Instrument to assess anxiety severity. The HAM-A was one of the first rating scales developed to measure the severity of anxiety symptoms. The scale consists of 14 items, each defined by a series of symptoms, and measures both psychic anxiety (mental agitation and psychological distress) and somatic anxiety (physical complaints related to anxiety). Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe. It was administered by a clinician experienced in working with psychiatric patients.
Hamilton Depression Scale (HAM-D) | 0-4-12 weeks
  Otherwise known as Hamilton Rating Scale for Depression or HRSD-17. The patient is rated by a clinician on 21 items scored either on a 3-point or 5-point Likert-type scale. Although the form lists 21 items, the scoring is based on the first 17. It generally takes 15-20 minutes to complete the interview and score the results. Eight items are scored on a 5-point scale, ranging from 0 = not present to 4 = severe. Nine are scored from 0-2. A score of 0-7 is considered to be normal while a score of 20 or higher indicates at least moderate severity.
20-Item Toronto Alexithymia Scale (TAS-20) | 0-4-12 weeks
  Instrument to assess alexithymia severity. The TAS is a 20-item instrument with 3 subscales: 1) difficulty Describing Feelings subscale, is used to measure difficulty describing emotions. 5 items; 2) difficulty Identifying Feeling subscale is used to measure difficulty identifying emotions. 7 items; 3) Externally-Oriented Thinking subscale, is used to measure the tendency of individuals to focus their attention externally. 8 items. The scale is a self-report scale that is comprised of 20 items. Items are rated using a 5-point Likert scale whereby 1 = strongly disagree and 5 = strongly agree. There are 5 items that are negatively keyed (items 4, 5, 10, 18 and 19). The total alexithymia score is the sum of responses to all 20 items, while the score for each subscale factor is the sum of the responses to that subscale. The TAS-20 uses cutoff scoring: equal to or less than 51 = non-alexithymia, equal to or greater than 61 = alexithymia. Scores of 52 to 60 = possible alexithymia.
Coping Orientation to the Problems Experienced (COPE-NIV) | 0-4-12 weeks
  instrument for measuring a broad range of coping styles

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Paolucci, MD, PhD, Principal Investigator — Università "Sapienza" Roma
Locations (1):
- Umberto I Hospital, Rome, Italy